CLINICAL TRIAL: NCT02484755
Title: Targeted Therapy With Gefitinib in Patients With USP8-mutated Cushing's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, associate professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2015-167
Record Dates: First submitted 2015-06-21; First posted 2015-06-30 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Cushing's Disease; Corticotrophin Adenoma
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gefitinib (Experimental): gifitinib 250 mg oral administration once daily for a total of 4 weeks.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — See Arm Description

SUMMARY:
The USP8 gene and its downstream target, epidermal growth factor receptor (EGFR), is a potential therapeutic target of Cushing disease. The EGFR inhibitor, Gefitinib, has been shown to reduce the production of ACTH both in vitro and in vivo, especially in USP8-mutated corticotrophin adenomas. The investigators hypothesize that Gefitinib will suppress pituitary corticotroph tumor ACTH production and normalize urinary free cortisol levels in patients with USP8-mutated Cushing's disease. Gefitinib is an FDA approved drug used to treat non-small cell lung cancer. However, in this study, the drug will be used to treat corticotrophin adenoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or greater
* Patients with confirmed diagnosis of ACTH-dependent Cushing's disease as evidenced by

  * Mean urinary free cortisol of four 24-hour urine samples collected within 2 weeks, at least 1.5 times the upper limit of the laboratory normal range
  * Morning plasma ACTH within the normal or above normal range
  * Either MRI confirmation of pituitary macroadenoma (greater than or equal to 1 cm), or inferior petrosal sinus gradient >3 after CRH stimulation for those patients with a microadenoma (tumor less than 1 cm)*, or for patients who have had prior pituitary surgery, histopathology confirming an ACTH staining adenoma.

    * if IPSS had previously been performed without CRH (e.g.with DDAVP), then a central to peripheral pre-stimulation gradient > 2 is required. If IPSS had not previously been performed, IPSS with CRH stimulation is required.
* Patients with de novo Cushing's disease can be included only if they are not considered candidates for pituitary surgery (e.g. poor surgical candidates, surgically unapproachable tumors, patients who refuse to have surgical treatment)
* Confirmatory testing prior to IPSS (low-dose dexamethasone suppression testing or dexamethasone-CRH testing) has to be performed for patients with UFC ≤ 3.0 X ULN and a pituitary microadenoma in order to exclude possible pseudo-Cushing's syndrome.
* Karnofsky performance status ≥ 60 (i.e. requires occasional assistance, but is able to care for most of this personal needs)
* For patients on medical treatment for Cushing's disease the following washout periods must be completed before baseline efficacy assessments are performed

  * Inhibitors of steroidogenesis (ketoconazole, metyrapone, rosiglitazone): 1 week
  * Dopamine agonists (bromocriptine, cabergoline): 4 weeks
  * Octreotide LAR and Lanreotide autogel: 8 weeks
  * Lanreotide SR: 4 weeks
  * Octreotide (immediate release formulation): 1 week
* Patients with a known history of impaired fasting glucose or DM may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary

Exclusion Criteria:

* Patients who have received pituitary irradiation within the last ten years prior to visit 1, as the onset time of the radiation effects cannot be determined
* Patients who have treated with mitotane during the last 6 months prior to Visit 1
* Patients with compression of the optic chiasm causing any visual field defect, in order to exclude patients with a tumor causing chiasma compression requiring surgery
* Patients with Cushing's syndrome due to ectopic ACTH secretion
* Patients with hypercortisolism secondary to adrenal tumors or nodular (primary) bilateral adrenal hyperplasia
* Patients who have a known inherited syndrome as the cause for hormone over secretion (i.e. Carney Complex, McCune-Albright syndrome, MEN-1)
* Patients with a diagnosis of glucocorticoid-remedial aldosteronism (GRA)
* Patients who are hypothyroid and not on adequate replacement therapy
* Patients who have undergone major surgery within 1 month prior to starting the study
* Patients with symptomatic cholelithiasis
* Diabetic patients on antidiabetic medications whose fasting blood glucose is poorly controlled as evidenced by HbA1C >8%
* Patients with abnormal coagulation (PT or PTT elevated by 30% above normal limits)
* Patients receiving anticoagulants that affect PT or PTT
* Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, advanced heart block, history of acute MI less than one year prior to study entry or clinically significant impairment in cardiovascular function
* Patients with risk factors for torsade de pointes, i.e. patients with a baseline QTc >480 ms, hypokalemia, family history of long QT syndrome, and concomitant medications known to prolong QT interval
* Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with ALT/AST more than 2 X ULN, serum creatinine >2.0 X ULN, serum bilirubin >2.0 X ULN, serum albumin < 0.67 X LLN
* Patients with WBC <3 X 109/L; Hgb < LLN; PLT <100 X 109/L
* Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results in the opinion of the investigator or the sponsor's medical monitor
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method for birth control. Female patients must use barrier contraception with condoms. If oral contraception is used, the patient must have been practicing this method for at least two months prior to enrollment and must agree to continue the oral contraceptive throughout the course of the study and for one month after the last dose of study drug. Male patients who are sexually active are required to use condoms during the study and for 1 month afterwards
* History of immunocompromise, including a positive HIV test result (Elisa and Western blot). An HIV test will not be required, however, previous medical history will be reviewed
* Patients who have a history of alcohol or drug abuse in the 6 month period prior to receiving pasireotide
* Patients who have given a blood donation (of 400 ml or more) within 2 months before receiving gefitinib
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to dosing and patients who have previously been treated with gefitinib
* Known hypersensitivity to gefitinib
* Patients with active malignant disease within the last five years (with the exception of basal cell carcinoma or carcinoma in situ of the cervix)
* Patients with the presence of active or suspected acute or chronic uncontrolled infection
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in levels of 24 hour urinary free cortisol after 4 weeks | Baseline, Week 4
  Full response is defined as the reduction of 24 hour urinary free cortisol more than 50% or normalized. Partial response is defined as the reduction of 24 hour urinary free cortisol between 25%~ 50%. Poor response or resistance is defined as the reduction of 24 hour urinary free cortisol less than 25%.

SECONDARY OUTCOMES:
Number of participants with a normalized 24 hour urinary free cortisol after 4 weeks | 4 weeks
Change in levels of Late-Night Salivary Cortisol after 4 weeks | Baseline, Week 4
Change in levels of pituitary hormones （a composite of pituitary panel) | Baseline, Week 4
  Pituitary Panel (TSH,FT4, FT3, PRL, IGF-1, FSH, Testosterone Total, Free Testosterone, Estradial, SHBG)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 weeks
Changes in tumor size | Baseline, Week 4
Changes in clinical signs (the typical signs of Cushing's Disease such as facial rubor, hirsutism, striae, bruising and supraclavicular and dorsal fat pad) | Baseline, Week 4
  The following symptoms will be evaluated using photographs taken at baseline and at the end of the study (Week 4):
  facial rubor, hirsutism, striae, bruising and supraclavicular and dorsal fat pad. The photographs will be assessed (scored) by the investigator as well as a second qualified physician at the site, who is blinded to the timepoint at which the photographs were taken.

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, MD, Principal Investigator — Department of Neurosurgery, Huashan Hospital, Fudan University
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China